CLINICAL TRIAL: NCT03054350
Title: Phase 2, Randomized, Double-Blind, Placebo Controlled, Dose-Finding Study to Assess the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Vadadustat in Japanese Subjects With Anemia Secondary to Dialysis-Dependent Chronic Kidney Disease (DD-CKD)
Brief Title: Dose-Finding Study of Vadadustat in Japanese Subjects With Anemia Secondary to Dialysis-Dependent Chronic Kidney Disease (DD-CKD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0022
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Anemia; Dialysis Dependent Chronic Kidney Disease
Keywords: Anemia; kidney; dialysis dependent chronic kidney disease; CKD; DD; renal; vadadustat; AKB-6548; hypoxia-inducible factor; Akebia (AKB); hypoxia-inducible factor (HIF); HIF; prolyl-hydroxylase inhibitor (PHI); PHI; Japan; Japanese
MeSH Terms: conditions — Anemia | interventions — vadadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | US Export: Yes

ARMS (4):
- Vadadustat, Dose 1 (Experimental): Daily oral dose
  Interventions: Drug: Vadadustat
- Vadadustat, Dose 2 (Experimental): Daily oral dose
  Interventions: Drug: Vadadustat
- Vadadustat, Dose 3 (Experimental): Daily oral dose
  Interventions: Drug: Vadadustat
- Placebo (Placebo Comparator): Daily oral dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vadadustat — Daily oral dose
  Other Names: AKB-6548
  Arms: Vadadustat, Dose 1; Vadadustat, Dose 2; Vadadustat, Dose 3
Drug: Placebo — Daily oral dose
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, dose-finding study to assess the efficacy, safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) of orally administered vadadustat in Japanese participants with anemia secondary to Dialysis-dependent Chronic Kidney Disease (DD-CKD).

ELIGIBILITY:
Inclusion Criteria:

* Male and female Japanese participants ≥20 years of age
* Receiving chronic maintenance hemodialysis for end-stage kidney disease
* Hemoglobin (Hb) <10.0 grams per deciliter (g/dL)

Exclusion Criteria:

* Anemia due to a cause other than chronic kidney disease (CKD) or presence of active bleeding or recent blood loss
* Sickle cell disease, myelodysplastic syndromes, bone marrow fibrosis, hematologic malignancy, myeloma, hemolytic anemia, thalassemia, or pure red cell aplasia
* Red blood cell transfusion within 4 weeks prior to or during screening
* Anticipated to recover adequate kidney function to no longer require hemodialysis during study participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2018-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (18):
- Japan (18):
  - Aichi
  - Ehime
  - Fukui
  - Hiroshima
  - Hokkaido
  - Hyōgo
  - Ibaraki
  - Kagoshima
  - Kochi
  - Miyagi
  - Nagano
  - Nagasaki
  - Niigata
  - Okinawa
  - Osaka
  - Ōita
  - Saitama
  - Shizuoka

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had not recently received erythropoiesis-stimulating agent (ESA) therapy participated in 2 screening visits (SVs). Participants who had recently received ESA therapy and otherwise met the eligibility criteria were required to washout from ESA therapy prior to evaluation of screening hemoglobin levels and participate in 3 SVs.
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 milligrams (mg), administered as 1 tablet once daily (QD), for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target hemoglobin (Hb) of 10.0 to 12.0 grams/deciliter (g/dL) based on dose adjustment guidelines.
- Vadadustat 300 mg: Participants were randomized to receive vadadustat 300 mg, administered as 2 tablets QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Vadadustat 600 mg: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Placebo to Vadadustat 150 mg: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 150 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Placebo to Vadadustat 300 mg: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 300 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Placebo to Vadadustat 600 mg: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 600 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
Period: Primary Efficacy Period (6 Weeks)
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Started | 15 | 15 | 15 | 5 | 5 | 5
Completed | 11 | 13 | 13 | 3 | 1 | 2
Not Completed | 4 | 2 | 2 | 2 | 4 | 3
Not completed — ESA Rescue/Blood Transfusion for Anemia | 4 | 2 | 1 | 2 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Dose Adjustment and Maintenance Period
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Started | 11 | 13 | 13 | 3 | 1 | 2
Completed | 10 | 13 | 12 | 2 | 1 | 2
Not Completed | 1 | 0 | 1 | 1 | 0 | 0
Not completed — ESA Rescue/Blood Transfusion for Anemia | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Captured as Other | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Population, comprised of all enrolled participants who received at least 1 dose of study medication. The Safety Population was based on the actual treatment that participants received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg | Total
Number analyzed (Participants) | 15 | 15 | 15 | 5 | 5 | 5 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.01) | 64.3 (8.02) | 65.1 (9.05) | 60.8 (12.85) | 61.0 (15.60) | 70.8 (8.23) | 63.8 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 5 | 2 | 3 | 2 | 19
  Male | 10 | 13 | 10 | 3 | 2 | 3 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hemoglobin Levels [Mean (Standard Deviation); unit: grams per deciliter (g/dL)] — Population: Data are reported for members of the Modified Intent-to-Treat (mITT) Population, comprised of all randomized participants who received at least 1 dose of study medication, had a pre-treatment Hb average, and at least one post-Baseline Hb measurement. The mITT Population was based on the treatment to which participants were randomized.
  grams per deciliter (g/dL)
    number analyzed (Participants) | 15 | 15 | 14 | 5 | 4 | 5 | 58
    (all) | 8.996 (0.5229) | 8.793 (0.5254) | 9.317 (0.6222) | 8.827 (0.6405) | 8.950 (0.7331) | 9.133 (0.6737) | 9.015 (0.5935)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin (Hb) Levels From Pre-treatment to the End of the Primary Efficacy Period
Description: The pre-treatment average value for Hb was defined as the average of 3 values obtained prior to treatment, i.e., the qualifying screening value and the Baseline value. Change from Pre-treatment was calculated as the Week 6 value minus the Pre-treatment value.
Time Frame: Pre-treatment; Week 6
Population: Modified Intent-to-Treat Population (mITT): all randomized participants who received at least 1 dose of study medication, had a pre-treatment Hb average, and at least one post-Baseline Hb measurement. The mITT Population was based on the treatment to which participants were randomized.
Measure: Least Squares Mean (Standard Error); unit: grams per deciliter (g/dL)
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 milligrams (mg), administered as 1 tablet once daily (QD), for 6 weeks.
- Vadadustat 300 mg: Participants were randomized to receive vadadustat 300 mg, administered as 2 tablets QD, for 6 weeks.
- Vadadustat 600 mg: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets QD, for 6 weeks.
- Placebo: Participants were randomized to receive matching placebo for 6 weeks.
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 14
grams per deciliter (g/dL) | -0.28 (0.218) | 0.08 (0.222) | 0.41 (0.233) | -1.48 (0.226)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Test type: Superiority; p = 0.0004, ANCOVA; The analysis of covariance (ANCOVA) model includes treatment assignment (3 dosed groups; 1 placebo group) and pre-treatment Hb value as a covariate; Least squares mean difference = 1.19, 95% CI 2-sided [0.56 to 1.82], Standard Error of Mean 0.314
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model includes treatment assignment (3 dosed groups; 1 placebo group) and pre-treatment Hb value as a covariate; Least squares mean difference = 1.56, 95% CI 2-sided [0.93 to 2.19], Standard Error of Mean 0.315
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 2]; Least squares mean difference = 1.89, 95% CI 2-sided [1.23 to 2.54], Standard Error of Mean 0.326

2. Secondary Outcome: Time to Reach the Target Hb Level of 10.0 to 12.0 g/dL From Baseline up to Week 16
Description: Time for this analysis was measured from Day 1 (Baseline) through the point in time during either the Primary Efficacy Period or the Dose Adjustment and Maintenance Period when a participant's Hb level achieved the target range of 10.0 to 12.0 g/dL.
Time Frame: from Baseline up to Week 16
Population: mITT Population. Only participants with Hb < 10.0 g/dL at the Baseline visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target hemoglobin (Hb) of 10.0 to 12.0 grams/deciliter (g/dL) based on dose adjustment guidelines.
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 8 | 12 | 11 | 0 | 2 | 1
days | 69.3 (25.31) | 79.2 (24.94) | 54.6 (27.90) |  | 57.0 (19.80) | 85.0 (NA) — A standard deviation was not calculated for a single participant.

3. Secondary Outcome: Mean Hb Levels at the End of the Primary Efficacy Period
Description: Data are reported as mean of the actual Week 6 values.
Time Frame: up to Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet once daily QD, for 6 weeks.
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 11 | 13 | 13 | 6
g/dL | 9.064 (1.0652) | 9.062 (0.8412) | 9.969 (0.7296) | 7.817 (1.4662)

4. Secondary Outcome: Mean Hb Levels at the End of the Dose Adjustment and Maintenance Period
Description: Data are reported as mean of the actual Week 16 values.
Time Frame: up to Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet OD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Vadadustat 300 mg: Participants were randomized to receive vadadustat 300 mg, administered as 2 tablets OD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Vadadustat 600 mg: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets OD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 10 | 13 | 12 | 2 | 1 | 2
g/dL | 10.460 (0.7501) | 11.285 (1.7841) | 11.100 (1.1402) | 8.600 (0.9899) | 13.200 (NA) — A standard deviation was not calculated for a single participant. | 12.100 (1.5556)

5. Secondary Outcome: Number of Participants Who Achieved the Target Hb Level of 10.0 to 12.0 g/dL at the End of the Dose Adjustment and Maintenance Period
Time Frame: up to Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 10 | 13 | 12 | 2 | 1 | 2
Participants | 7 | 11 | 7 | 0 | 0 | 1

6. Secondary Outcome: Mean Change in Hb Between Pre-treatment and the End of the Dose Adjustment and Maintenance Period
Description: A pre-treatment average value for Hb was defined as the average of 3 values obtained prior to dosing, i.e., the 2 qualifying screening values and the Baseline value. Change from Pre-treatment was calculated as the Week 16 value minus the Pre-treatment value.
Time Frame: Pre-treatment; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 10 | 13 | 12 | 2 | 1 | 2
g/dL | 1.397 (0.5755) | 2.444 (1.7807) | 1.644 (1.4973) | -0.233 (0.1414) | 3.800 (NA) — A standard deviation was not calculated for a single participant. | 3.000 (0.2828)

7. Secondary Outcome: Mean Change in Red Blood Cell (RBC) Count and Absolute Reticulocyte Count From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: 10^6 cells/microliter (µL)
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet QD, for 6 weeks.
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 11 | 13 | 13 | 6
10^6 cells/microliter (µL)
  RBC Count | -0.01 (0.073) | 0.08 (0.069) | 0.20 (0.069) | -0.30 (0.099)
  Absolute Reticulocyte Count | 0.02 (0.005) | 0.02 (0.004) | 0.03 (0.004) | 0.01 (0.006)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; RBC Count; Test type: Superiority; p = 0.0232, ANCOVA; The ANCOVA model will include treatment assignment (3 dosed groups;1 placebo group) and pre-treatment Hb value as a covariate; Least squares mean difference = 0.29, 95% CI 2-sided [0.04 to 0.54], Standard Error of Mean 0.122
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; RBC Count; Test type: Superiority; p = 0.0033, ANCOVA; The ANCOVA model will include treatment assignment (3 dosed groups; 1 placebo group) and pre-treatment Hb value as a covariate; Least squares mean difference = 0.38, 95% CI 2-sided [0.13 to 0.62], Standard Error of Mean 0.121
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; RBC Count; Test type: Superiority; p = 0.0002, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 0.50, 95% CI 2-sided [0.26 to 0.74], Standard Error of Mean 0.120
Statistical Analysis 4: Comparison: Vadadustat 150 mg vs Placebo; Absolute Reticulocyte Count; Test type: Superiority; p = 0.3289, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 0.01, 94% CI 2-sided [-0.01 to 0.02], Standard Error of Mean 0.008
Statistical Analysis 5: Comparison: Vadadustat 300 mg vs Placebo; Absolute Reticulocyte Count; Test type: Superiority; p = 0.2607, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 0.01, 95% CI 2-sided [-0.01 to 0.02], Standard Error of Mean 0.007
Statistical Analysis 6: Comparison: Vadadustat 600 mg vs Placebo; Absolute Reticulocyte Count; Test type: Superiority; p = 0.0252, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 0.02, 95% CI 2-sided [0.00 to 0.03], Standard Error of Mean 0.007

8. Secondary Outcome: Mean Change in RBC Count and Absolute Reticulocyte Count From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^6 cells/µL
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 10 | 13 | 12 | 2 | 1 | 2
10^6 cells/µL
  RBC Count | 0.454 (0.2225) | 0.819 (0.5127) | 0.503 (0.5056) | 0.065 (0.0212) | 1.160 (NA) — A standard deviation was not calculated for a single participant. | 1.035 (0.0778)
  Absolute Reticulocyte Count | 0.017 (0.0169) | 0.021 (0.0180) | 0.016 (0.0162) | 0.016 (0.0083) | 0.024 (NA) — A standard deviation was not calculated for a single participant. | 0.014 (0.0217)

9. Secondary Outcome: Mean Change in Hematocrit and Reticulocytes From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 11 | 13 | 13 | 6
percentage
  Hematocrit | 0.67 (0.770) | 1.98 (0.737) | 3.30 (0.737) | -2.63 (1.045)
  Reticulocytes | 0.64 (0.158) | 0.57 (0.141) | 0.71 (0.140) | 0.39 (0.212)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Hematocrit; Test type: Superiority; p = 0.0154, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 3.31, 95% CI 2-sided [0.67 to 5.94], Standard Error of Mean 1.303
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Hematocrit; Test type: Superiority; p = 0.0008, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 4.61, 95% CI 2-sided [2.06 to 7.16], Standard Error of Mean 1.261
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Hematocrit; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 5.93, 95% CI 2-sided [3.31 to 8.56], Standard Error of Mean 1.296
Statistical Analysis 4: Comparison: Vadadustat 150 mg vs Placebo; Reticulocytes; Test type: Superiority; p = 0.3572, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 0.25, 95% CI 2-sided [-0.30 to 0.81], Standard Error of Mean 0.273
Statistical Analysis 5: Comparison: Vadadustat 300 mg vs Placebo; Reticulocytes; Test type: Superiority; p = 0.4758, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 0.18, 95% CI 2-sided [-0.33 to 0.69], Standard Error of Mean 0.252
Statistical Analysis 6: Comparison: Vadadustat 600 mg vs Placebo; Reticulocytes; Test type: Superiority; p = 0.2048, ANCOVA; [statistical method as in outcome 7, analysis 2]; Least squares mean difference = 0.33, 95% CI 2-sided [-0.19 to 0.84], Standard Error of Mean 0.254

10. Secondary Outcome: Mean Change in Hematocrit and Reticulocytes From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 10 | 13 | 12 | 2 | 1 | 2
percentage
  Hematocrit | 5.12 (2.105) | 8.92 (5.100) | 5.63 (4.921) | 1.20 (0.000) | 12.90 (NA) — A standard deviation was not calculated for a single participant. | 10.70 (1.697)
  Reticulocytes | 0.32 (0.636) | 0.33 (0.686) | 0.24 (0.547) | 0.55 (0.212) | 0.40 (NA) — A standard deviation was not calculated for a single participant. | 0.15 (0.636)

11. Secondary Outcome: Mean Change in Iron and Total Iron Binding Capacity (TIBC) From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms per deciliter (μg/dL)
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 11 | 13 | 13 | 6
micrograms per deciliter (μg/dL)
  Iron | -3.3 (26.60) | -1.5 (19.50) | -8.1 (21.95) | -1.5 (26.64)
  TIBC | 35.4 (28.72) | 67.5 (25.72) | 80.7 (39.04) | 15.8 (8.08)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Iron; Test type: Superiority; p = 0.9373, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Iron; Test type: Superiority; p = 0.6623, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Iron; Test type: Superiority; p = 0.9374, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 4: Comparison: Vadadustat 150 mg vs Placebo; TIBC; Test type: Superiority; p = 0.2085, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 5: Comparison: Vadadustat 300 mg vs Placebo; TIBC; Test type: Superiority; p = 0.0016, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 6: Comparison: Vadadustat 600 mg vs Placebo; TIBC; Test type: Superiority; p = 0.0001, ANCOVA; test of treatment group difference based on ANCOVA model

12. Secondary Outcome: Mean Change in Iron and TIBC From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 10 | 13 | 12 | 2 | 1 | 2
μg/dL
  Iron | -18.5 (24.01) | -8.7 (24.29) | 0.9 (48.22) | -9.5 (30.41) | -7.0 (NA) — A standard deviation was not calculated for a single participant. | 15.0 (43.84)
  TIBC | 58.5 (44.12) | 80.9 (29.42) | 85.4 (39.91) | 33.0 (2.83) | 108.0 (NA) — A standard deviation was not calculated for a single participant. | 78.0 (62.23)

13. Secondary Outcome: Mean Change in Transferrin Saturation (TSAT) From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 11 | 13 | 13 | 6
percentage | -6.51 (11.621) | -10.14 (11.294) | -12.46 (9.544) | -2.78 (12.822)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Test type: Superiority; p = 0.2708, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Test type: Superiority; p = 0.0966, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Test type: Superiority; p = 0.0424, ANCOVA; test of treatment group difference based on ANCOVA model

14. Secondary Outcome: Mean Change in TSAT From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 10 | 13 | 12 | 2 | 1 | 2
percentage | -14.25 (12.069) | -13.79 (13.549) | -10.93 (12.627) | -12.50 (18.526) | -17.10 (NA) — A standard deviation was not calculated for a single participant. | -4.70 (12.021)

15. Secondary Outcome: Mean Change in Ferritin and Hepcidin From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 11 | 13 | 13 | 6
nanograms per milliliter (ng/mL)
  Ferritin | -51.20 (58.855) | -68.67 (54.707) | -104.49 (49.558) | 12.63 (32.424)
  Hepcidin | -53.465 (43.5531) | -73.587 (32.3547) | -104.301 (36.7636) | -11.802 (13.6518)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Ferritin; Test type: Superiority; p = 0.0207, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Ferritin; Test type: Superiority; p = 0.0022, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Ferritin; Test type: Superiority; p < 0.0001, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 4: Comparison: Vadadustat 150 mg vs Placebo; Hepcidin; Test type: Superiority; p = 0.0062, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 5: Comparison: Vadadustat 300 mg vs Placebo; Hepcidin; Test type: Superiority; p = 0.0002, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 6: Comparison: Vadadustat 600 mg vs Placebo; Hepcidin; Test type: Superiority; p < 0.0001, ANCOVA — test of treatment group difference based on ANCOVA model

16. Secondary Outcome: Mean Change in Ferritin and Hepcidin From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 10 | 13 | 12 | 2 | 1 | 2
ng/mL
  Ferritin | -105.09 (55.837) | -119.28 (84.000) | -113.52 (54.559) | -43.05 (81.954) | -150.70 (NA) — A standard deviation was not calculated for a single participant. | -76.95 (42.356)
  Hepcidin | -73.826 (50.9042) | -99.367 (51.3174) | -106.838 (40.1472) | -95.940 (98.7262) | -122.300 (NA) — A standard deviation was not calculated for a single participant. | -35.140 (62.9184)

17. Secondary Outcome: Number of Participants Who Required Rescue With a RBC Transfusion From Baseline to the End of the Primary Efficacy Period
Description: Participants who initiated rescue therapy (including RBC transfusion) were required to stop study drug treatment and were discontinued from the study.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 14
Participants | 0 | 0 | 1 | 3

18. Secondary Outcome: Number of Participants Who Required Rescue With RBC Transfusion From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: as for outcome 17
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 15 | 15 | 14 | 5 | 4 | 5
Participants | 1 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants Who Required Rescue With Erythropoiesis-Stimulating Agents (ESAs) From Baseline to the End of the Primary Efficacy Period
Description: ESA rescue is defined as participants with ESA administration and 1) the participant experienced a clinically significant worsening of their anemia or symptoms of anemia, 2) the participant's Hb level is <9.0 g/dL, and 3) reason for early study withdrawal of worsening of anemia requiring ESA rescue or blood transfusion. Participants who initiated rescue therapy (including ESAs) were required to stop study drug treatment and were discontinued from the study.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 14
Participants | 4 | 2 | 1 | 8

20. Secondary Outcome: Number of Participants Who Required Rescue With ESAs From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: as for outcome 19
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 15 | 15 | 14 | 5 | 4 | 5
Participants | 0 | 0 | 0 | 1 | 0 | 0

21. Secondary Outcome: Number of the Participants With the Indicated Number of Dose Adjustments From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Increases in dose were not allowed during the 6-week Primary Efficacy Period.
Time Frame: up to Week 16
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 15 | 15 | 14 | 5 | 4 | 5
Participants
  0 dose adjustments | 5 | 3 | 9 | 2 | 3 | 3
  1 dose adjustment | 2 | 2 | 2 | 1 | 0 | 0
  2 dose adjustments | 5 | 8 | 3 | 1 | 1 | 2
  3 or more dose adjustments | 3 | 2 | 0 | 1 | 0 | 0

22. Secondary Outcome: Plasma Concentration Profile of Vadadustat and Its Metabolites Using a Pre-dose Sample From Week 4
Description: Blood samples were collected for analysis.
Time Frame: Week 4, pre-dose
Population: Pharmacokinetic (PK) Population: all participants in the Safety Population (all enrolled participants who received at least 1 dose of study medication) who had a pre-dose PK sample at Week 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 13 | 13 | 0
μg/mL
  Vadadustat | 4343.54 (175.17) | 7561.36 (134.77) | 15083.03 (46.77) |
  O-glucuronide | 8667.97 (73.79) | 14623.89 (67.44) | 36476.33 (57.18) |
  Acyl-glucuronide | 12.019 (16.55) | 12.174 (8.10) | 22.765 (70.53) |

23. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (SAEs) in the Primary Efficacy Period
Description: An adverse event (AE) was defined as any untoward medical occurrence (including a clinically significant abnormal laboratory finding) that occurred in the protocol-specified AE reporting period. An AE included medical conditions, signs, and symptoms not previously observed in the participant that emerged during the protocol-specified AE reporting period, including signs or symptoms associated with pre-existing underlying conditions that were not present prior to the AE reporting period. An AE that met one or more of the following criteria or outcomes was classified as serious: death; life-threatening; in-patient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; was considered a medically important event not meeting the above criteria, but which could jeopardize a participant, or could require medical or surgical intervention to prevent one of the criteria listed in this definition.
Time Frame: up to Week 6
Population: Safety Population: all enrolled participants who received at least 1 dose of study medication. The Safety Population was based on the actual treatment that participants received
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  TEAEs | 8 | 11 | 6 | 6
  Treatment-emergent SAEs | 0 | 0 | 3 | 1

24. Secondary Outcome: Number of Participants With TEAEs and Treatment-emergent SAEs in the Dose Adjustment and Maintenance Period
Description: An AE was defined as any untoward medical occurrence (including a clinically significant abnormal laboratory finding) that occurred in the protocol-specified AE reporting period. An AE included medical conditions, signs, and symptoms not previously observed in the participant that emerged during the protocol-specified AE reporting period, including signs or symptoms associated with pre-existing underlying conditions that were not present prior to the AE reporting period. An AE that met one or more of the following criteria or outcomes was classified as serious: death; life-threatening; in-patient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; was considered a medically important event not meeting the above criteria, but which could jeopardize a participant, or could require medical or surgical intervention to prevent one of the criteria listed in this definition.
Time Frame: up to Week 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 15 | 15 | 15 | 5 | 5 | 5
Participants
  TEAEs | 9 | 9 | 9 | 1 | 1 | 2
  Treatment-emergent SAEs | 1 | 1 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to Week 18
Groups:
- Primary Efficacy Period: 150 mg Vadadustat: Participants were randomized to receive vadadustat 150 milligrams (mg), administered as 1 tablet once daily (QD), for 6 weeks.
- Primary Efficacy Period: 300 mg Vadadustat: Participants were randomized to receive vadadustat 300 mg, administered as 2 tablets QD, for 6 weeks.
- Primary Efficacy Period: 600 mg Vadadustat: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets QD, for 6 weeks.
- Primary Efficacy Period: Placebo Matched to 150 mg Vadadustat; Primary Efficacy Period: Placebo Matched to 300 mg Vadadustat; Primary Efficacy Period: Placebo Matched to 600 mg Vadadustat: Participants were randomized to receive matching placebo for 6 weeks.
- Dose Adjustment and Maintenance: 150 mg Vadadustat: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target hemoglobin (Hb) of 10.0 to 12.0 grams/deciliter (g/dL) based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: 300 mg Vadadustat: Participants were randomized to receive vadadustat 300 mg, administered as 2 tablets QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: 600 mg Vadadustat: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: Placebo to 150 mg Vadadustat: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period.
  During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 150 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: Placebo to 300 mg Vadadustat: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period.
  During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 300 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: Placebo to 600 mg Vadadustat: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period.
  During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 600 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
Arm/Group | Primary Efficacy Period: 150 mg Vadadustat | Primary Efficacy Period: 300 mg Vadadustat | Primary Efficacy Period: 600 mg Vadadustat | Primary Efficacy Period: Placebo Matched to 150 mg Vadadustat | Primary Efficacy Period: Placebo Matched to 300 mg Vadadustat | Primary Efficacy Period: Placebo Matched to 600 mg Vadadustat | Dose Adjustment and Maintenance: 150 mg Vadadustat | Dose Adjustment and Maintenance: 300 mg Vadadustat | Dose Adjustment and Maintenance: 600 mg Vadadustat | Dose Adjustment and Maintenance: Placebo to 150 mg Vadadustat | Dose Adjustment and Maintenance: Placebo to 300 mg Vadadustat | Dose Adjustment and Maintenance: Placebo to 600 mg Vadadustat
All-Cause Mortality (participants affected / at risk) | 8/15 | 11/15 | 6/15 | 2/5 | 2/5 | 2/5 | 9/15 | 9/15 | 9/15 | 1/5 | 1/5 | 2/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 3/15 | 0/5 | 1/5 | 0/5 | 1/15 | 1/15 | 1/15 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 8/15 | 11/15 | 5/15 | 2/5 | 2/5 | 2/5 | 9/15 | 9/15 | 9/15 | 1/5 | 1/5 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Efficacy Period: 150 mg Vadadustat (N=15) | Primary Efficacy Period: 300 mg Vadadustat (N=15) | Primary Efficacy Period: 600 mg Vadadustat (N=15) | Primary Efficacy Period: Placebo Matched to 150 mg Vadadustat (N=5) | Primary Efficacy Period: Placebo Matched to 300 mg Vadadustat (N=5) | Primary Efficacy Period: Placebo Matched to 600 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: 150 mg Vadadustat (N=15) | Dose Adjustment and Maintenance: 300 mg Vadadustat (N=15) | Dose Adjustment and Maintenance: 600 mg Vadadustat (N=15) | Dose Adjustment and Maintenance: Placebo to 150 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: Placebo to 300 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: Placebo to 600 mg Vadadustat (N=5)
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Efficacy Period: 150 mg Vadadustat (N=15) | Primary Efficacy Period: 300 mg Vadadustat (N=15) | Primary Efficacy Period: 600 mg Vadadustat (N=15) | Primary Efficacy Period: Placebo Matched to 150 mg Vadadustat (N=5) | Primary Efficacy Period: Placebo Matched to 300 mg Vadadustat (N=5) | Primary Efficacy Period: Placebo Matched to 600 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: 150 mg Vadadustat (N=15) | Dose Adjustment and Maintenance: 300 mg Vadadustat (N=15) | Dose Adjustment and Maintenance: 600 mg Vadadustat (N=15) | Dose Adjustment and Maintenance: Placebo to 150 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: Placebo to 300 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: Placebo to 600 mg Vadadustat (N=5)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 5 | 1 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site erosion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular graft stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT03054350/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT03054350/SAP_001.pdf